## Official title:

This study was part of Beijing Osteoporosis with Neurological Disorders in Epigenetic Changes Study (BONE)

## **NCT** number:

NCT03401619

## **Document date**

15<sup>th</sup> September, 2020

Peking University Third Hospital, Peking University

BONE study is a community-based and ambispective cohort study of clinical and subclinical osteoporosis with neurological disorders disease. Between 2017 and 2018, BONE study enrolled 2,000 adults aged 55-102 from six communities in Beijing district (Mu dan yuan community, Ji men li community, Xiao nan zhuang community, Lan qi ying community, Jiu xian qiao community, Chang chun jie community).

## **Statistical Analysis Plan**

Continuous variables are described as mean (standard deviation), and categorical variables are described as frequency (percentage). Student's t test was used to evaluate the difference of continuous variables, and Pearson's  $\chi 2$  test or Fisher's exact test was used to evaluate the difference of categorical variables. We used Cox proportional hazards models with age as the timescale to assess the relationship between residential proximity to major roadways and the incidence of osteoporotic fracture.

For each outcome, follow up time (in days) was measured from Sept 27, 2007 until osteoporotic fracture date, or Sept 26, 2017. Separate models were developed for osteoporotic fracture. All models were adjusted for age, household economic status, education, physical activity, diet, smoking, alcohol, comorbidities and Risk factors for osteoporotic fractures. Two co-authors perform statistical analysis and cross-check to ensure quality. SPSS (version 17.0; IBM, Inc) is used for all statistical analysis. Two-sided P values of less than 0.05 were considered statistically significant.